CLINICAL TRIAL: NCT00732927
Title: Parnaparin Versus Aspirin in the Treatment of Retinal Vein Occlusion. A Randomized, Double Blind, Controlled Study
Brief Title: Parnaparin vs Aspirin in the Treatment of Retinal Vein Occlusion
Acronym: PARVO
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: slow recruitment rate
Sponsor: Università degli Studi dell'Insubria (Other)
Collaborators: Alfa Wassermann, Bologna, Italy (Unknown)
Responsible Party: Walter Ageno, University of Insubria
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: FLU/OVR/001/2001
Record Dates: First submitted 2008-08-07; First posted 2008-08-12 (Estimated); Last update posted 2008-08-12 (Estimated); Status verified 2008-08

CONDITIONS: Retinal Vein Occlusion
Keywords: thrombosis, vein, retina
MeSH Terms: conditions — Retinal Vein Occlusion; Thrombosis | interventions — parnaparin; Aspirin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): parnaparin, low molecular weight heparin
  Interventions: Drug: parnaparin
- 2 (Active Comparator): aspirin
  Interventions: Drug: aspirin

INTERVENTIONS:
Drug: parnaparin — vials, 6.400 IU sc twice daily for 7 days, then once daily for a total of 3 months
  Arms: 1
Drug: aspirin — tablets, 100 mg for 3 months
  Arms: 2

SUMMARY:
Retinal vein occlusion (RVO) is the second commonest retinal disease after diabetic retinopathy, and is a common cause of unilateral visual loss. There are two aims in the management of RVO: the identification of modifiable risk factors and their medical management and the recognition and management of sight-threatening complications. The management of the disease includes laser therapy and the control of systemic associated diseases. Many other treatments have been proposed but there is no evidence on their efficacy in modulating the outcome of branch or central RVO. There are currently no adequate clinical trials that have evaluated the efficacy and safety of antithrombotic agents in this setting. Antiplatelet agents are frequently used in clinical practice. Anticoagulant drugs, either heparins or coumarins, are also used in this setting as they represent the first line therapy for the treatment of venous thromboembolism. Aim of this randomized controlled study is to to compare the efficacy and safety of aspirin and of a low molecular weight heparin, parnaparin, in the treatment of RVO. Study treatment is administered for 3 months. Primary end-point of the study is the incidence of functional worsening of the eye with RVO at 6 months. Secondary efficacy outcomes are the following: proportion of cases requiring laser treatment because of the extension of the ischemic lesion and/or the presence of neovascularisation and/or macular oedema, incidence of recurrent RVO objectively documented by fluorescein angiography. Safety outcomes are defined by the incidence of major and minor bleeding events.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 85 years
* A body weight of greater than 50 Kg
* A requirement that no more than 15 days had passed between symptomatic presentation, confirmation of RVO and entry into the study.

Exclusion Criteria:

* Modification of the optic media transparency that could compromise the evaluation of fluorescein angiography, such as cataract or corneal degeneration
* History of major ocular surgery (with the exclusion of cataract extraction)
* Previous RVO
* Other ocular conditions that, in the opinion of the investigator, could have affected macular edema or altered visual acuity during the course of the study - Contraindications to the study drugs (e.g. major bleeding or neurosurgical procedures in the previous 3 months, serum creatinine levels of greater than 2.0 mg/dL, severe liver insufficiency, platelet count < 100,000 mm3, known active peptic gastric ulcer)
* Active malignancy
* Pregnancy
* Inability to attend for follow up or anticipated non-compliance
* Ongoing treatment with aspirin or anticoagulant drugs at the time of RVO diagnosis

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2002-07; Primary Completion 2006-07 (Actual); Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
incidence of functional worsening of the eye with RVO | 6 months

SECONDARY OUTCOMES:
proportion of cases requiring laser treatment | 6 months
incidence of recurrent RVO | 6 months
incidence of major and minor bleeding events | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Davide Imberti, MD, Study Director — Ospedale di Piacenza; Roberto Cattaneo, MD, Study Director — Ospedale di Gallarate; Walter Ageno, MD, Study Chair — Università degli Studi dell'Insubria
Locations (1):
- University Of Insubria, Varese, Italy

REFERENCES:
- [Derived] Ageno W, Cattaneo R, Manfredi E, Chelazzi P, Venco L, Ghirarduzzi A, Cimino L, Filippucci E, Ricci AL, Romanelli D, Incorvaia C, D'Angelo S, Campana F, Molfino F, Scannapieco G, Rubbi F, Imberti D. Parnaparin versus aspirin in the treatment of retinal vein occlusion. A randomized, double blind, controlled study. Thromb Res. 2010 Feb;125(2):137-41. doi: 10.1016/j.thromres.2009.05.007. Epub 2009 May 27. PMID 19477488